CLINICAL TRIAL: NCT02781168
Title: Influence of the Use of Hearing Protection in the Salivary Cortisol Level and in the Sleep of Premature Infants: Clinical, Randomized, Controlled, Crossover
Brief Title: Influence of the Use of Hearing Protection in the Salivary Cortisol Level and in the Sleep of Premature Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Mavilde da Luz Gonçalves Pedreira, Teacher, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UFSP 2
Record Dates: First submitted 2016-05-09; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Premature Newborn
Keywords: Premature newborn; Cortisol; Stress
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Use of earmuffs (Experimental): The earmuffs are brand Natus® Pediatrics, Neonatal Noise Attenuators called MiniMuffs®, San Carlos, California, USA, which allow the reduction of sound pressure levels 7 to 12 decibels.
  Interventions: Device: use of earmuffs
- No use of earmuffs (Active Comparator): No use of earmuffs are brand Natus® Pediatrics, Neonatal Noise Attenuators called MiniMuffs®, San Carlos, California, USA, which allow the reduction of sound pressure levels 7 to 12 decibels.
  Interventions: Device: use of earmuffs

INTERVENTIONS:
Device: use of earmuffs — The earmuffs are brand Natus® Pediatrics, Neonatal Noise Attenuators called MiniMuffs®, San Carlos, California, USA, which allow the reduction of sound pressure levels 7 to 12 decibels. Are devices that have oval and anatomical shape that allow proper positioning of the ears of newborns. They are made with a soft foam and has hydrogel adhesive on the outer edges for attachment to the skin.

SUMMARY:
The aim of this study was to investigate the influence of the use of headphones in salivary cortisol levels in newborns (NB) during periods of nap aimed at noise reduction, brightness and handling NB, measure the concentrations of salivary cortisol before (baseline) and after the use of hearing protection (response) in the neonatal intensive care unit (NICU).

A NICU nap periods and compare the influence of the use and non-use of hearing protection in salivary cortisol levels and sleep patterns of infants during nap periods of the NICU.

DETAILED DESCRIPTION:
The aim of this study was to investigate the influence of the use of headphones in salivary cortisol levels in newborns (NB) during periods of nap aimed at noise reduction, brightness and handling NB, measure the concentrations of salivary cortisol before (baseline) and after the use of hearing protection (response) in the NICU nap periods and compare the influence of the use and non-use of hearing protection in salivary cortisol levels and sleep patterns of infants during nap periods of the NICU. Being the chance prosposta the use of headphones during periods of environmental control has an influence on the level of salivary cortisol and sleep in preterm infants.

This is a randomized clinical trial, controlled, crossover, in which clinical intervention is introduced by the researcher that controls and varies, featuring experimental research.

In this study the intervention being tested is the use of hearing protection in infants. The ear is employed in certain periods of the day. These periods established by the Neonatal Intensive Care Unit (ICU), are intended to promote environmental noise control and manipulation of the NB.

Levels of cortisol present in the saliva of the newborn will be analyzed, allowing to measure the biologically active free cortisol in the body.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn male or female;
* Inside the incubator;
* Clinically stable;
* No change in evoked otoacoustic emissions;
* Current weight between 1200 to 2000g.

Exclusion Criteria:

* In phototherapy;
* In invasive mechanical ventilation and noninvasive;
* With any type of congenital malformation;
* Periventricular hemorrhage with grade II, III and IV;
* In using any medication depressant, analgesic or corticosteroid in last 24 hours;
* Premature newborn whose mother has a history of illicit drug use during pregnancy.

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of Salivary Cortisol Levels and the Use of Hearing Protection | 19 months
  The aim of this study was to investigate the influence of the use of earmuffs in salivary cortisol levels in newborns (NB) during periods of nap aimed at noise reduction.
Sleep of premature infants and use of earmuffs | 19 months
  The aim of this study was to investigate the influence of the use of earmuffs in the sleep in premature infants.

CONTACTS AND LOCATIONS:
Overall Officials: Mavilde LG Pedreira, PhD, Principal Investigator — Federal University of São Paulo; Fabricia M Araujo, RN, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No